CLINICAL TRIAL: NCT01979250
Title: Fuchs' Endothelial Dystrophy: Clinical Characteristics, Treatment Outcome, and Pathology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Esben Nielsen, MD, Aarhus University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSAEKtrial1
Record Dates: First submitted 2013-10-30; First posted 2013-11-08 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Fuchs' Endothelial Corneal Dystrophy
Keywords: endothelial keratoplasty; Descemet's stripping automated endothelial keratoplasty; lamellar keratoplasty
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy | interventions — Descemet Stripping Endothelial Keratoplasty; Corneal Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal corneas (No Intervention): Normal corneas from patients that undergo cataract surgery.
- DSAEK surgery (Other): Corneal endothelial transplantation by Descemet's stripping automated endothelial keratoplasty (DSAEK).
  Interventions: Procedure: DSAEK surgery

INTERVENTIONS:
Procedure: DSAEK surgery — Corneal endothelial transplantation by "Descemet's stripping automated endothelial keratoplasty" (DSAEK).
  Other Names: DSEK; Endothelial keratoplasty; Lamellar keratoplasty; Descemet's stripping automated endothelial keratoplasty
  Arms: DSAEK surgery

SUMMARY:
Background Fuchs' Endothelial Dystrophy Fuchs' Endothelial Dystrophy (Fuchs' ED) is characterized by changes on the inside of the cornea, which leads to a substantial decline in visual acuity. The only effective treatment option for Fuchs' ED is corneal transplantation.

Corneal transplantation Corneal transplantation surgery has seen major advances in the last decade, and the Descemet's Stripping Automated Endothelial Keratoplasty (DSAEK) procedure has now become the preferred method.

Outcome There have been a substantial number of publications on outcome after DSAEK surgery, and the procedure has several advantages over the former preferred method of transplantation, penetrating keratoplasty (PK).

Despite the apparent success of the DSAEK procedure, visual acuity is seldom fully restored even in otherwise healthy eyes. Several studies have tried to clarify this matter but so far results have been conflicting.

Hypotheses

1. The reduction in visual acuity and contrast sensitivity in patients with Fuchs' endothelial dystrophy is correlated with corneal thickness, corneal light scatter, and the type and magnitude of optical disrupting guttae in Descemet's membrane.
2. The subjective visual function after corneal transplantation with a posterior lamellar graft is correlated with the optical properties of the grafted cornea (thickness, light scatter, irregularities on the anterior, and posterior corneal surfaces)

Materials and methods

In a controlled prospective trial of DSAEK patients, we aim to register different morphological patterns, monitor visual performance and optical parameters.

Three sex and age-matched groups will be compared:

Group 1: 40 patients that undergo DSAEK surgery Group 2: 40 patients that undergo combined cataract and DSAEK surgery. Group 3: Control group of 40 patients with normal corneas that undergo cataract surgery.

DETAILED DESCRIPTION:
Investigation outline:

* Presence of the following patterns will be registered for each patient: Scattered guttae, confluent guttae, diffuse corneal oedema or confined corneal oedema
* Refractive properties: Objective and subjective refraction
* Visual performance: Visual acuity (ETDRS), Contrast sensitivity (FrACT method)
* Corneal characterization: corneal sensibility (Cochet-Bonnet), In vivo confocal microscopy, specular microscopy, anterior segment OCT, OLCR, Pentacam with densitometry, and slit-lamp investigation will be performed.
* Catquest 9SF questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Fuchs' endothelial dystrophy
* Candidate for DSAEK surgery

Exclusion Criteria:

* other ocular comorbidities that potentially limit vision or contrast vision

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2013-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Visual acuity | Up to 3 years

OTHER OUTCOMES:
Refractive properties, corneal clarity, subjective satisfaction | Up to 3 years
  Subjective satisfaction will be measured using the Catquest 9SF questionnaire which uses a Likert scale which in turn is converted into a Rasch scale. The scales is linear, and uses a unit called the logit.

CONTACTS AND LOCATIONS:
Overall Officials: Esben Nielsen, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Department of Ophthalmology, Aarhus, Aarhus C, Denmark

REFERENCES:
- [Result] Nielsen E, Ivarsen A, Kristensen S, Hjortdal J. Fuchs' endothelial corneal dystrophy: a controlled prospective study on visual recovery after endothelial keratoplasty. Acta Ophthalmol. 2016 Dec;94(8):780-787. doi: 10.1111/aos.13126. Epub 2016 Jun 7. PMID 27273977
- Available data/document: Manuscript — http://www.ncbi.nlm.nih.gov/pubmed/27273977 — To acces the results, please go to the above mentioned manuscript.